CLINICAL TRIAL: NCT03834922
Title: PROMPT Providing Standardized Consented PROMs (Patient Reported Outcome Measures) for Improving Pain Treatment A Multicenter, Non-interventional, Prospective Observational Study
Brief Title: Providing Standardized Consented PROMs (Patient Reported Outcome Measures) for Improving Pain Treatment
Acronym: PROMPT
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Winfried Meissner (Other)
Collaborators: Grünenthal GmbH (Industry); University Hospital Muenster (Other); Hospital Ambroise Paré Paris (Other); Novartis Pharmaceuticals (Industry); Hôpital Raymond Poincaré (Other); University of Helsinki (Other); University Hospital St Luc, Brussels (Other); Oxford University Hospitals NHS Trust (Other); University Hospital, Geneva (Other); Orthopedic Center Santy, Lyon, France (Unknown); University of Naples (Other); Hospital Clínico Universitario de Valladolid (Other); Cancer Center Porto, Portugal (Unknown); Orthopedic Institute Banjika, Belgrade, Serbia (Unknown); Cardiovascular Center Dedinje, Belgrade, Serbia (Unknown); University of Homburg (Other); Barts & The London NHS Trust (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital Dresden (Other); University Hospital Bergmannsheil Bochum (Other); Infirmerie Protestante de Lyon (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Winfried Meissner, Study coordinator, University of Jena
Organization: University of Jena (Other)
Other Study IDs: 777500-IMI-PainCare PROMPT
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative
Keywords: Acute pain; Chronification of pain; Pain treatment; Pain management; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Total knee arthroplasty: Patients undergoing total knee arthroplasty
  Interventions: Other: Prospective data collection
- Sternotomy: Patients undergoing sternotomy
  Interventions: Other: Prospective data collection
- Breast: Patients undergoing breast surgery
  Interventions: Other: Prospective data collection
- Endometriosis: Patients undergoing endometriosis-related surgery
  Interventions: Other: Prospective data collection

INTERVENTIONS:
Other: Prospective data collection — No intervention. It's a prospective data collection.

SUMMARY:
PROMPT aims at improving management of acute and chronic pain by identifying a core set of PROMs (patient reported outcome measures) that are predictive indicators of treatment success in clinical practice and controlled trials. These will not only address pain intensities as well as the functional consequences of pain for individuals but also identify patients at risk of experiencing chronification of acute post-operative pain. Results will help health care professionals to individualize pain management, and thus improve the quality of life of pain patients.

DETAILED DESCRIPTION:
In order to reach this objective, a non-interventional prospective data collection aiming at reaching a consensus on a core set of PROMs which reliably predict and/or measure success in acute and chronic pain treatments in real life conditions and identifying predictors for chronification of postoperative pain will be conducted (PROMPT NIT-1). Aim of the data collection is to evaluate the abilities of certain PROMs in assessing acute post-surgical pain outcomes in daily routine care of patients after four different surgical procedures: (total knee replacement, breast surgery, sternotomy and surgery related to endometriosis), and to validate selected risk factors for chronification prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of consenting age (>18 years old)
* Elective surgery
* Planned stay in hospital for the surgery
* First contact with the patient before surgery
* Patient agrees to participate

Exclusion Criteria:

* Patient is unable to give consent
* Cognitive impairment
* Questionnaire is not available in a language the patient is fluent in
* Patient not willing to answer the follow-up questionnaire

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — For the groups 'Breast' and 'Endometriosis', only female patients can be included.
Study Population: Patients undergoing one of the following types of surgery: TKA, breast, sternotomy and endometriosis related surgery. Only female patients will be included in the Breast Surgery and Endometriosis group. For the other surgeries, there will not be a special preference in the distribution by sex or age for the recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 3322 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
WP 2 - Acute pain: Sensitivity to change | 2019 - 2022
  For WP2, the primary endpoint will be pain intensity at day 3 (NRS Scale from 0 to 10, 0 being no pain, 10 being worst pain imaginable). This primary endpoint (PROMs) will be used to assess sensitivity to change from POD3 to POD1.
WP 3 - Chronification of pain: Incidence of chronic post-surgical pain (CPSP) | 2019 - 2022
  For WP3, the primary end point will be the incidence of moderate to severe CPSP (Numeric rating scale ≥ 3/10) at 6 months using the average pain on the Brief Pain Inventory Questionnaire.

SECONDARY OUTCOMES:
Objective physical activity and sleep, measured with Actigraph devices | 01/2020 to 12/2021
  Correlation of physical activity data (average no. of steps of days 5 to 7) with PRO "physical function" on day 7;
Association between other POD7 PROMs and activity/sleep | 01/2020 to 12/2021
  Association between other POD7 PROMs and activity/sleep
Association between peri-operative processes and activity/sleep | 01/2020 to 12/2021
  Association between peri-operative processes and activity/sleep
Is decreased activity a predictor for chronic postsurgical pain? | 01/2020 to 12/2021
  Is decreased activity a predictor for chronic postsurgical pain on POM6?
Do activity trajectories since surgery parallel trajectories of other outcomes? | 01/2020 to 12/2021
  Do activity trajectories since surgery parallel trajectories of other outcomes?
Correlation of activity difference between POD5-7 and preop with POD7 oucomes | 01/2020 to 12/2021
  Correlation of activity difference between POD5-7 and preop with POD7 oucomes
Association between ambient light intensity and outcomes on POD7 | 01/2020 to 12/2021
  Association between ambient light intensity and outcomes on POD7

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Meissner, Prof., Study Chair — Jena University Hospital; Hiltrud Liedgens, Dr., Study Chair — Grünenthal GmbH; Esther Pogatzki-Zahn, Prof., Principal Investigator — University Hospital Münster; Dominique Fletcher, Prof., Principal Investigator — Hospital Ambroise Paré Paris; Shaloo Pandhi, Principal Investigator — Novartis
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vollert J, Egert VM, Segelcke D, Fletcher D, Kalso E, Kemp H, Lavand'homme P, Komann M, Weinmann C, Meissner W, Pogatzki-Zahn EM. Minimal Clinically Important Changes of Patient-reported Outcome Measures for Acute Postsurgical Pain. Anesthesiology. 2026 Jan 1;144(1):143-153. doi: 10.1097/ALN.0000000000005792. Epub 2025 Oct 9. PMID 41065659
- [Derived] Martinez V, Lehman T, Lavand'homme P, Harkouk H, Kalso E, Pogatzki-Zahn EM, Komann M, Meissner W, Weinmann C, Fletcher D. Chronic postsurgical pain: A European survey. Eur J Anaesthesiol. 2024 May 1;41(5):351-362. doi: 10.1097/EJA.0000000000001974. Epub 2024 Feb 27. PMID 38414426